CLINICAL TRIAL: NCT00849355
Title: Phase II, Multicenter Trial to Evaluate the Efficacy and Safety of the Following Treatment Squeme:Ciclophosphamide, Vincristine, Lyposomal Doxorrubicine, Myocet and Prednisone,Combined With Rituximab in First Line Treatment for Patients With Aggresive No Hodgkin B Lymphoma and Cardiovascular Risk
Brief Title: Ciclophosphamide, Vincristine, Myocet and Prednisone, With Rituximab in 1st-Line Treatment for Patients With No-Hodgkin B Lymphoma and Cardiovascular (CV) Risk
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asociacion Doctor Peset Para el Estudio de la Hematología (Other)
Collaborators: Cephalon (Industry); Pivotal S.L. (Industry)
Responsible Party: Secundino Ferrer, Asociacion Doctor Peset Para el Estudio de la Hematología
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADOPEH-LINFMYO-2007
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2009-02-23 (Estimated); Status verified 2009-02

CONDITIONS: No Hodgkin B Lymphoma
MeSH Terms: interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- unique (Experimental): RCOMP-14 with Rituximab
  Interventions: Drug: RCOMP-14 + rituximab

INTERVENTIONS:
Drug: RCOMP-14 + rituximab — Pretreatment: vincristine 1mg at day -6 and Methylprednisolone 100 mg from -6 to day 0.
  Treatment: rituximab 375m/m2 + ciclophosphamide 750 mg/m2 + Vincristine 1.4 mg/m2 + Doxorrubicine 50 mg/m2 at day 1 and every 14d. Prednisone 100 mg/d from day 1 to 5 and every 14 d.

SUMMARY:
The purpose of this study is to evaluate the efficacy (and safety) of the following treatment squeme:Ciclophosphamide, Vincristine, lyposomal Doxorrubicine (Myocet) and Prednisone,combined with Rituximab in first line treatment for patients with aggresive No Hodgkin B lymphoma and cardiovascular risk

DETAILED DESCRIPTION:
Phase II, multicenter, open , 1-arm study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological diagnosis of Lymphoma no Hodgkin B CD20+ high degree of mailgnancy
2. Patients no previously treated
3. stage III o IV
4. Informed consent
5. At least one measurable injury
6. Age >18
7. ECOG 0-2
8. Life expectancy >6 months
9. Cardiovascular risk defined as:Mild-moderate systolic dysfunction,isquemic cardiopathy, diabetes mellitus, hypertension,left ventricular hypertrophy, cardiac arrhythmia, moderate pulmonar hypertension
10. adequate organic functionallity (creatinine<2mg/dl;bilirubin<2mg/dl; ALT-AST-FA<5 FSN; neutrphyls total count >1.5x 109/l and platellet count >100x1097l)
11. Use of a contraceptive method during study + 3 months -

Exclusion Criteria:

1. stage I or II with IPI=0
2. Symptomatic tumoral affection of Nervous central system
3. Lymphoma no hodgkin B indolent
4. Lymphoma no hodgkin B mantle-cell
5. Lymphoma no hodgkin T
6. lymphoprolifertaive syndrome post-transplantation or immunosuppression associated
7. cardiovacualr disease symptomatic
8. Cronic infection or acute serious
9. history of neoplasia in past 5 years
10. not able to understand the study or poor protocol adherence
11. Known Hypersensivity to any atudy drug
12. pregnant/lactant women
13. Previous participation in clinicla study in past 30 days
14. Previous treatment with antraciclines or any drug used in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate treatment efficacy by measuring response to treatment | at the end of study

SECONDARY OUTCOMES:
evaluate cardiotoxicity and tolerability | At the end of study
Evaluate progression free survival | At the end of study
Evaluate event free survival | At the end of study
Evaluate tumor free survival | At the end of study
Evaluate overall survival | At the end of study
Evaluate response duration | At the end of study
treatment adherence | At the end of study
time to progression | At the end of the study
dose intensity and relative dose intensity | At the end of the study

CONTACTS AND LOCATIONS:
Locations (12):
- Spain (12):
  - hospital del Mar, Barcelona
  - Hospital Vall D'Hebrón, Barcelona
  - Hospital de Castellon, Castellon
  - Hospital Severo Ochoa, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital de Getafe, Madrid
  - Hospital son Llatzer, Mallorca
  - Hospital Morales Messeguer, Murcia
  - Hospital Santa Mª del Rosell, Murcia
  - Hospital general universitario de Valencia, Valencia
  - H. Arnau de Vilanova, Valencia
  - Hospital Universitario Dr. Peset, Valencia